CLINICAL TRIAL: NCT07186790
Title: Risk Factors for Initial Non Invasive Ventilation Failure in Preterms With Gestational Age <32 Weeks in Neonatal Intensive Care Units of Assiut University Children Hospital ,One Year Study
Brief Title: Non-invasive Ventilation
Acronym: CPAP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara mohamed hadia mohamed, Principal investigator, Assiut University
Other Study IDs: Non invasive ventilation
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Non Invasive Ventilation Failure in Preterms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Risk factors for non invasive ventilation failure in preterms that lead them to use invasive ventilation

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is widely utilized in the initial respiratory management of very low birth weight (VLBW) preterms , particularly those born at a gestational age of less than 32 weeks, to avoid complications associated with invasive mechanical ventilation. Despite advances in neonatal respiratory care, the risk of initial NIV failure remains a significant clinical concern due to its association with increased morbidity and the subsequent need for intubation and invasive support. Early identification of neonates at high risk for NIV failure is crucial for timely intervention and optimization of respiratory strategies to improve outcomes (Wu et al., 2024).

Previous multicenter and prospective studies have highlighted various clinical and physiological parameters contributing to the failure of NIV in preterms. These include lower gestational age, severe respiratory distress syndrome (RDS), higher oxygen requirements, and hemodynamic instability in the immediate postnatal period (Boix et al., 2023). The complexity of respiratory adaptation in this population necessitates robust risk stratification tools and predictive models to support clinical decision-making in the neonatal intensive care unit (NICU) (Fernandez-Gonzalez et al., 2022).

Recent research efforts, including the establishment of predictive models, have focused on incorporating variables such as Apgar scores, initial FiO₂, surfactant administration, and radiographic findings to identify preterms most likely to fail NIV. Understanding these risk factors is essential not only for improving survival but also for reducing the incidence of bronchopulmonary dysplasia (BPD) and other long-term pulmonary complications (Shen et al., 2024).

Furthermore, expert consensus guidelines from neonatology societies advocate for early use of continuous positive airway pressure (CPAP) and targeted surfactant therapy to mitigate the progression of RDS and enhance NIV success. However, despite adherence to best practices, a considerable proportion of VLBW preterms still experience respiratory deterioration necessitating escalation to invasive ventilation (Akin et al., 2025).

Emerging data also point to institution-specific practices, such as type of NIV modality used (e.g., nasal intermittent positive pressure ventilation vs. high-frequency oscillatory NIV) (Wang et al., 2025).

Given the significant clinical implications, understanding and applying these risk factors can help neonatal teams anticipate NIV failure early, apply targeted respiratory strategies, and improve short- and long-term outcomes in preterms (Afzal et al., 2024; de Souza Júnior et al., 2023; Yazici et al., 2025).

ELIGIBILITY:
Inclusion Criteria:

-

The study will include neonates who meet all of the following criteria:

1. Preterms born at a gestational age of less than 32 weeks.
2. Birth weight less than 1,500 grams (very low birth weight).
3. Received initial non-invasive ventilation (e.g., CPAP or HFNC) within the first hours of life.
4. Admitted to participating NICUs during the study period.
5. Complete medical records available for review and analysis.

Exclusion Criteria:

-

Preterms will be excluded from the study if they meet any of the following conditions:

1. Received immediate invasive mechanical ventilation at birth without a trial of non-invasive ventilation.
2. Presence of major congenital anomalies (e.g., congenital diaphragmatic hernia, significant cardiac malformations).
3. Diagnosed with chromosomal abnormalities or genetic syndromes.
4. Incomplete or missing medical records that prevent accurate data extraction.
5. Preterms transferred from another hospital after initiation of respiratory support.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of preterms aged <32 weeks and what is the risk factors for failure of non invasive ventilation that lead them to use invasive ventilation
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Risk factors for initial non invasive ventilation failure in preterms with gestational age <32 weeks in neonatal intensive care units of assiut university children hospital,one year study | One year
  Risk factors for initial non invasive ventilation failure in preterms with gestational age <32 weeks in neonatal intensive care units of assiut university children hospital,one year study

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bastos de Souza Junior NW, Rosa TR, Cerantola JCK, Ferrari LSL, Probst VS, Felcar JM. Predictive factors for extubation success in very low and extremely low birth weight preterm infants. Can J Respir Ther. 2023 Sep 15;59:204-213. doi: 10.29390/001c.87789. eCollection 2023. PMID 37781349
- [Background] Fernandez-Gonzalez SM, Sucasas Alonso A, Ogando Martinez A, Avila-Alvarez A. Incidence, Predictors and Outcomes of Noninvasive Ventilation Failure in Very Preterm Infants. Children (Basel). 2022 Mar 17;9(3):426. doi: 10.3390/children9030426. PMID 35327798
- [Background] Yazici A, Buyuktiryaki M, Sari FN, Alyamac Dizdar E. Risk factors for noninvasive ventilation failure in preterm infants at less than 30 weeks of gestation with respiratory distress syndrome. J Trop Pediatr. 2024 Dec 5;71(1):fmae051. doi: 10.1093/tropej/fmae051. PMID 39840596
- [Background] Wang W, Tan R, Dong W. Non-invasive intermittent positive pressure ventilation vs non-invasive high-frequency oscillatory ventilation as post-extubation support in extremely birth weight infants: a retrospective study. Eur J Pediatr. 2025 Apr 21;184(5):303. doi: 10.1007/s00431-025-06117-5. PMID 40257605
- [Background] Shen F, Yu MY, Rong H, Guo Y, Zou YS, Cheng R, Yang Y. Establishment and Validation of a Risk Prediction Model for Non-Invasive Ventilation Failure After Birth in Premature Infants with Gestational Age < 32 Weeks. Lung. 2024 Oct;202(5):543-552. doi: 10.1007/s00408-024-00727-w. Epub 2024 Jul 3. PMID 38958717
- [Background] Akin MS, Sari FN, Cetinkaya AK, Acikgoz IC, Dizdar EA. The Predictors and Outcomes of Early Noninvasive Positive Pressure Ventilation Failure in Very Preterm Infants: A Prospective Study. Am J Perinatol. 2025 Jun 16. doi: 10.1055/a-2624-5642. Online ahead of print. PMID 40523391